CLINICAL TRIAL: NCT05776186
Title: Fetal Heart Rate Pattern Before, During, and After Spinal Anesthesia for Scheduled Uncomplicated Cesarean Section
Brief Title: Fetal Heart Rate Pattern After Spinal Anesthesia for Scheduled Uncomplicated Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CF22379A
Record Dates: First submitted 2022-12-02; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Continuous Fetal Heart Beat Monitor and Analysis After Spinal Anesthesia
Keywords: cesarean section; spinal anesthesia ; fetal heart beat
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before spinal anesthesia: Before spinal anesthesia with heavy bupivacaine 12.5 mg is administrated.
  Interventions: Drug: Spinal anesthesia with heavy bupivacaine
- After spinal anesthesia: After spinal anesthesia with heavy bupivacaine 12.5 mg is administrated.
  Interventions: Drug: Spinal anesthesia with heavy bupivacaine

INTERVENTIONS:
Drug: Spinal anesthesia with heavy bupivacaine — Spinal anesthesia

SUMMARY:
Spinal anesthesia may cause sympathetic blockade which decrease peripheral vascular resistance and bradycardia and then hypotension. Maternal hypotension could cause immediate fetus heart beat (FHB) deceleration and postpartum acidosis. Both intravenous hydration or vasopressor during hypotension could prevent maternal hypotension efficiently. Although there were many articles discussion about maternal hypotension and fetal heart rate variation during epidural labor analgesia, the studies about FHB variation during spinal anesthesia is not much. In one literature in 1960, if maternal blood pressure below 60-80 mmHg, FHB deceleration could happen in 5 minutes. In modern medical management, FHB change during and after spinal anesthesia is an interesting topic. The most relevant study was published by NTUH in 2015, which transformed EKG signal to possible FHB change.

The parturient will have FHB recording for 20 minutes in the day before operation. On the operation day, after proper position by the anesthetic staff (lateral position or sitting position), spinal anesthesia will performed by obstetric anesthesiologist and the lying down for supine position. Before the baby was delivered by cesarean section no FHB will be monitored. The aim of the study is continuous FHB monitor and analysis after spinal anesthesia for 5-10 minutes to improve fetal physiology knowledge and providing basic information for future study.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 20 years
2. Singleton
3. Gestational age above 36 weeks
4. Scheduled Cesarean section at VGHTC
5. Eligible for spinal anesthesia
6. Inform consent

Exclusion Criteria:

1. ASA > 3
2. Prenatal examination reveal suspect neonatal congenital heart disease, heart failure, arrythymia or hydrops fetalis which could affect fetal heart beat
3. Regular uterine contraction, premature rupture of membrane or vaginal bleeding before scheduled C/S on prenatal clinic
4. Anticipate vaginal delivery initially but shift to C/S for prolong labor, FHB deceleration or other reason
5. Patients cannot make decision for language barrier, education condition or phsycological disease
6. Register in other study already

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy women
Study Population: Pregnant women for gestational age above 36 weeks
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-10-13 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Fetal heart rate variability | 5 minutes after spinal anesthesia
  Fetal heart rate deceleration (normal > 100 beats per minute)

SECONDARY OUTCOMES:
Neonatal outcome | 1 minute and 5 minutes after delivery
  APGAR score_1 minute, APGAR score_5 minute ( APGAR score: 0-10 points)
Neonatal intensive care rate | baseline (admission)
  NICU admission rate
Umbilical vein analysis | within 5 minutes after delivery
  Umbilical vein blood gas analysis, including pH, O2, CO2, HgB, electrolyte
Maternal pain score | 0, 8, 24 hours after surgery
  Visual analog scale ( VAS score 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No